CLINICAL TRIAL: NCT01107912
Title: A Pharmacokinetic and Pharmacodynamic Comparison of Prasugrel and Clopidogrel in Very Elderly Versus Non-Elderly Aspirin-Treated Subjects With Stable Coronary Artery Disease
Brief Title: Comparison of Prasugrel and Clopidogrel in Very Elderly and Non-Elderly Patients With Stable Coronary Artery Disease
Acronym: GENERATIONS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12835; H7T-MC-TACY (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-09

CONDITIONS: Coronary Artery Disease
Keywords: Platelet function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 milligrams (mg) prasugrel (Experimental)
  Interventions: Drug: prasugrel
- 10 mg prasugrel (Active Comparator)
  Interventions: Drug: prasugrel
- 75 mg clopidogrel (Active Comparator)
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: prasugrel — administered orally, daily for 12 days
  Other Names: Efient; Effient; LY640315; CS747
  Arms: 10 mg prasugrel; 5 milligrams (mg) prasugrel
Drug: clopidogrel — Administered orally, daily for 12 days
  Arms: 75 mg clopidogrel

SUMMARY:
The 5-milligram (mg) maintenance dose (MD) of prasugrel in very elderly patients with coronary artery disease produces a pharmacodynamic response within the same therapeutic range as 10-mg MD in non-elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants (Either: at least 45 years of age, but less than 65 years of age OR 75 years of age or older) with a history of stable coronary artery disease who are not currently indicated for treatment with a thienopyridine (that is, prasugrel, clopidogrel, or ticlopidine)
* Provision of written informed consent
* Body weight greater than or equal to 60 kilograms (kg)
* For women of child-bearing potential only (that is, women who are not surgically or chemically sterilised and who are between menarche and 1 year post menopause), test negative for pregnancy (based on a urine or serum pregnancy test to be performed before randomisation) and agree to use a reliable method of birth control during the study

Exclusion Criteria:

* Unstable coronary artery disease
* Myocardial Infarction (MI) within the previous 30 days
* Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Graft Surgery (CABG) within the previous 90 days
* History of refractory ventricular arrhythmias within the last 6 months; an implanted defibrillator device; congestive heart failure within 6 months prior to screening; major surgery, or severe trauma, fracture or organ biopsy within 3 months prior to enrollment
* Any planned surgical procedure or any coronary revascularisation (surgical or percutaneous) planned within 60 days following randomisation
* Any known contraindication to treatment with an antiplatelet agent
* Significant hypertension at the time of screening or randomisation
* Clinically significant out-of-range values for platelet count or haemoglobin at screening, in the investigator's opinion, or results of clinical laboratory tests at the time of screening that are judged to be clinically significant for the study population, as determined by the investigator
* Prior history or presence of significant bleeding disorders, abnormal bleeding tendency, or personal history of coagulation or bleeding disorders
* Prior history or clinical suspicion of cerebral vascular malformations, intracranial neoplasm, Transient Ischemic Attack (TIA) or stroke
* Prior history of thrombocytopenia or thrombocytosis
* Use of antiplatelet agents (besides aspirin) within 10 days prior to screening; the use (or planned use) of heparin, oral anticoagulants, or fibrinolytic agents within 30 days of screening; or participants receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDS) or cyclooxygenase-2 (COX-2) inhibitors that cannot be discontinued for the duration of the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dublin, Ireland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nieuwegein, Netherlands
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo

REFERENCES:
- [Derived] Erlinge D, Gurbel PA, James S, Lindahl TL, Svensson P, Ten Berg JM, Foley DP, Wagner H, Brown PB, Luo J, Zhou C, Moser BA, Jakubowski JA, Small DS, Winters KJ, Angiolillo DJ. Prasugrel 5 mg in the very elderly attenuates platelet inhibition but maintains noninferiority to prasugrel 10 mg in nonelderly patients: the GENERATIONS trial, a pharmacodynamic and pharmacokinetic study in stable coronary artery disease patients. J Am Coll Cardiol. 2013 Aug 13;62(7):577-83. doi: 10.1016/j.jacc.2013.05.023. Epub 2013 Jun 7. PMID 23747759

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 mg Prasugrel (Elderly): Elderly participants (≥75 Years of Age) received 5 mg prasugrel for 12 days during Period 1 without intervening or terminal washout periods. They were then switched to either the 10 mg prasugrel or 75 mg clopidogrel dose in Period 2.
- 10 mg Prasugrel (Elderly): Elderly participants ( ≥75 year of age) on 5 mg prasugrel in Period 1 who received 10 mg prasugrel during Period 2 or 3.
- 75 mg Clopidogrel (Elderly): Elderly participants (≥75 year of age) on 5 mg prasugrel in Period 1 who received 75 mg clopidogrel during Period 2 or 3.
- 5 mg Prasugrel (Non-Elderly): Non-elderly participants (≥45 to <65 years of age) on 10 mg prasugrel in Period 1 who received 5 mg prasugrel during Period 2 or 3.
- 10 mg Prasugrel (Non-Elderly): Non-elderly participants (≥45 to <65 years of age) received 10 mg prasugrel for 12 days during Period 1 without intervening or terminal washout periods. They were then switched to either the 5 mg prasugrel or 75 mg clopidogrel dose in Period 2.
- 75 mg Clopidogrel (Non-Elderly): Non-elderly participants ( ≥45 to <65 years of age) on 10 mg prasugrel during Period 1 who received 75 mg clopidogrel during Period 2 or 3.
Period: Period 1
Arm/Group | 5 mg Prasugrel (Elderly) | 10 mg Prasugrel (Elderly) | 75 mg Clopidogrel (Elderly) | 5 mg Prasugrel (Non-Elderly) | 10 mg Prasugrel (Non-Elderly) | 75 mg Clopidogrel (Non-Elderly)
Started | 73 | 0 | 0 | 0 | 82 | 0
Received at Least 1 Dose of Study Drug | 73 | 0 | 0 | 0 | 82 | 0
Completed | 72 | 0 | 0 | 0 | 79 | 0
Not Completed | 1 | 0 | 0 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | 5 mg Prasugrel (Elderly) | 10 mg Prasugrel (Elderly) | 75 mg Clopidogrel (Elderly) | 5 mg Prasugrel (Non-Elderly) | 10 mg Prasugrel (Non-Elderly) | 75 mg Clopidogrel (Non-Elderly)
Started | 0 (Participants switched to either 10 mg prasugrel or 75 mg clopidogrel in Period 2.) | 36 | 36 | 41 | 0 (Participants switched to either 5 mg prasugrel or 75 mg clopidogrel in Period 2.) | 38
Completed | 0 | 36 | 35 | 41 | 0 | 38
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 3
Arm/Group | 5 mg Prasugrel (Elderly) | 10 mg Prasugrel (Elderly) | 75 mg Clopidogrel (Elderly) | 5 mg Prasugrel (Non-Elderly) | 10 mg Prasugrel (Non-Elderly) | 75 mg Clopidogrel (Non-Elderly)
Started | 0 | 35 (Participants who received 75 mg clopidogrel in Period 2 received 10 mg prasugrel in Period 3) | 36 (Participants who received 10 mg prasugrel in Period 2 received 75 mg clopidogrel in Period 3) | 38 (Participants who received 75 mg clopidogrel in Period 2 received 5 mg prasugrel in Period 3) | 0 | 41 (Participants who received 5 mg prasugrel in Period 2 received 75 mg clopidogrel in Period 3)
Completed | 0 | 34 | 35 | 37 | 0 | 41
Not Completed | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Very Elderly, Drug Sequence ABC: Participants (≥75 years of age) in this arm received study drug sequence ABC. A = Prasugrel 5mg, B = Prasugrel 10mg, C = Clopidogrel 75mg.
- Very Elderly; Drug Sequence ACB: Participants (≥75 years of age) in this arm received study drug sequence ACB. A = Prasugrel 5mg, B = Prasugrel 10mg, C = Clopidogrel 75mg.
- Non-Elderly; Drug Sequence BAC: Participants (≥45 to <65 years of age) in this arm received study drug sequence BAC. A = Prasugrel 5mg, B = Prasugrel 10mg, C = Clopidogrel 75mg.
- Non-Elderly; Drug Sequence BCA: Participants (≥45 to <65 years of age) in this arm received study drug sequence BCA. A = Prasugrel 5mg, B = Prasugrel 10mg, C = Clopidogrel 75mg.
- Total: Total of all reporting groups
Arm/Group | Very Elderly, Drug Sequence ABC | Very Elderly; Drug Sequence ACB | Non-Elderly; Drug Sequence BAC | Non-Elderly; Drug Sequence BCA | Total
Number analyzed (Participants) | 36 | 37 | 42 | 40 | 155
Age Continuous [Mean (Standard Deviation); unit: years] | 79.02 (2.87) | 78.74 (3.12) | 57.11 (4.75) | 55.46 (5.53) | 66.94 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 7 | 10 | 36
  Male | 28 | 26 | 35 | 30 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 7 | 9 | 14 | 38
  Unknown or Not Reported | 28 | 30 | 32 | 26 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 7 | 12
  White | 35 | 34 | 40 | 32 | 141
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 10 | 14 | 39
  Ireland | 3 | 3 | 7 | 6 | 19
  Netherlands | 3 | 4 | 2 | 1 | 10
  Sweden | 22 | 23 | 23 | 19 | 87
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 88.49 (10.92) | 82.30 (10.74) | 92.85 (20.01) | 93.36 (17.32) | 89.45 (16.01)
Tobacco Use Status at Baseline [Number; unit: participants]
  Yes | 4 | 1 | 13 | 11 | 29
  No | 32 | 36 | 29 | 29 | 126

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Platelet Aggregation (MPA) to 20 Micromoles (μM) Adenosine Diphosphate (ADP) as Measured by Light Transmission Aggregometry (LTA) From Baseline to 12 Days of Therapy in the First Treatment Period
Description: Maximum Platelet Aggregation (MPA) to 20 μM ADP was assessed by light transmission aggregometry (LTA), an assay that measures platelet aggregation by determining the amount of light transmitted through a cuvette containing the platelet-rich plasma stimulated with a platelet activator, such as ADP, relative to platelet-poor plasma (100% light transmittance). Lower MPA values reflect stronger platelet inhibition, whereas higher MPA values reflect weaker inhibition.
Time Frame: Baseline, 12 days
Population: All randomized participants who continued in the study through the Day 12 visit, and who had at least 1 evaluable PD assessment at the Day 12 visit. Participants were analysed based on randomized treatment assignment, regardless of the study drug they took.
Measure: Median (Inter-Quartile Range); unit: percentage of aggregation
Arm/Group | 5 mg Prasugrel (Elderly) | 10 mg Prasugrel (Non-Elderly)
Number analyzed (Participants) | 72 | 79
percentage of aggregation
  Baseline | 78.00 [72.00 to 83.50] | 75.00 [71.00 to 83.00]
  Period 1 (12 days) (n=71, 79) | 58.00 [50.00 to 65.00] | 46.00 [39.00 to 52.00]
Statistical Analysis 1: Comparison: 5 mg Prasugrel (Elderly) vs 10 mg Prasugrel (Non-Elderly); Test type: Non-Inferiority or Equivalence — The difference of median MPA to 20 μM ADP of a prasugrel 5-mg in the elderly group to the 75th percentile of the MPA to 20 μM ADP of a prasugrel 10 mg MD in the non-elderly group at the end of Period 1 was estimated from the observed data. The upper limit of the one-sided 97.5% confidence interval for the difference was estimated from resampling data with replacement through bootstrap methodology and was used to compare with the non-inferiority margin of 15 percentage points; Estimate of the difference = 6.00, 95% CI 2-sided [1.00 to 9.00]

2. Secondary Outcome: Change in Vasodilator-associated Stimulated Phosphoprotein (VASP) From Baseline to 12 Days of Therapy
Description: Vasodilator-associated stimulated phosphoprotein (VASP) phosphorylation levels, expressed as the platelet reactivity index (PRI), reflect the degree of thienopyridine-mediated P2Y12 receptor inhibition. A lower PRI reflects stronger inhibition of P2Y12, whereas a higher PRI reflects weaker inhibition of P2Y12.
Time Frame: Baseline, Day 12
Population: All randomized participants who received at least 1 dose of study drug and provided at least 1 evaluable pharmacodynamic (PD) measure at 1 of the 3 periods. Participants were analyzed based on the treatment they received for each period regardless of their randomized treatment assignment.
Measure: Mean (Standard Deviation); unit: percentage platelet reactive index (PRI)
Arm/Group | 5 mg Prasugrel (Elderly) | 10 mg Prasugrel (Elderly) | 75 mg Clopidogrel (Elderly) | 5 mg Prasugrel (Non-Elderly) | 10 mg Prasugrel (Non-Elderly) | 75 mg Clopidogrel (Non-Elderly)
Number analyzed (Participants) | 72 | 70 | 71 | 78 | 79 | 79
percentage platelet reactive index (PRI)
  Baseline (n=68, 66, 67, 71, 72, 72) | 85.62 (4.28) | 85.66 (4.32) | 85.60 (4.31) | 86.10 (5.31) | 86.18 (5.32) | 86.18 (5.32)
  Day 12 (n=67, 65, 67, 73, 74, 73) | 44.30 (18.87) | 22.66 (11.90) | 54.95 (18.86) | 54.72 (18.67) | 27.74 (15.84) | 54.53 (21.82)

3. Secondary Outcome: Change in VerifyNow P2Y12 Reaction Units (PRU) From Baseline to 12 Days of Therapy
Description: The Accumetrics VerifyNow® P2Y12 assay measures platelet aggregation in whole blood and is reported in P2Y12 reaction units (PRU). PRU report the extent of P2Y12 receptor-mediated platelet aggregation calculated as a function of the rate and extent of platelet aggregation in the presence of adenosine phosphate ADP. A lower PRU reflects stronger inhibition of P2Y12, whereas a higher PRU reflects weaker inhibition of P2Y12.
Time Frame: Baseline, Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: P2Y12 reaction units (PRU)
Arm/Group | 5 mg Prasugrel (Elderly) | 10 mg Prasugrel (Elderly) | 75 mg Clopidogrel (Elderly) | 5 mg Prasugrel (Non-Elderly) | 10 mg Prasugrel (Non-Elderly) | 75 mg Clopidogrel (Non-Elderly)
Number analyzed (Participants) | 72 | 70 | 71 | 78 | 79 | 79
P2Y12 reaction units (PRU)
  Baseline | 315.63 (45.98) | 314.11 (45.74) | 314.14 (44.54) | 291.81 (45.16) | 291.62 (44.90) | 291.62 (44.90)
  Day 12 (n=71, 67, 69, 77, 79, 79) | 175.52 (57.19) | 84.13 (47.72) | 212.33 (69.65) | 177.01 (67.29) | 85.46 (60.24) | 181.22 (71.80)

4. Secondary Outcome: Active Metabolite Blood Levels to Drug Exposure as Measured by Pharmacokinetics (PK) Through 4 Hours After Dosing
Description: A descriptive pharmacokinetic-pharmacodynamic (PK-PD) analysis comparing prasugrel and clopidogrel active metabolite exposures to MPA in response to 20 µM ADP (by LTA) was conducted as originally intended; however, the graphic output from that analysis is not possible here. Therefore, the PK portion is presented here as AUC and the PD portion is presented in Secondary Outcome Measure #5. AUC was calculated through the last scheduled sampling time of 4 hours [AUC (0-4)] or through the sampling time of the last quantifiable concentration prior to 4 hours. AUC values were denoted AUC(0-tlast) in both instances.
Time Frame: Baseline up to 4 hours post-dose
Population: All available PK sample data from all treated participants who contributed complete PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Units Other Than Participants: Participant PK Profiles
Arm/Group | 5 mg Prasugrel (Elderly) | 10 mg Prasugrel (Elderly) | 75 mg Clopidogrel (Elderly) | 5 mg Prasugrel (Non-Elderly) | 10 mg Prasugrel (Non-Elderly) | 75 mg Clopidogrel (Non-Elderly)
Number analyzed (Participants) | 71 | 70 | 70 | 78 | 80 | 79
Number analyzed (Participant PK Profiles) | 71 | 101 | 103 | 114 | 80 | 118
nanogram*hour/milliliter (ng*hr/mL) | 18.9 (43) | 41.2 (35) | 13.0 (62) | 16.1 (54) | 36.7 (49) | 11.8 (68)

5. Secondary Outcome: Change From Baseline in Maximum Platelet Aggregation (MPA) as Measured by Light Transmission Aggregometry (LTA) From Baseline at Day 12 of Therapy
Description: Maximum Platelet Aggregation (MPA) to 20 μM ADP was assessed by light transmission aggregometry (LTA), an assay that measures platelet aggregation by determining the amount of light transmitted through a cuvette containing the platelet-rich plasma stimulated with a platelet activator, such as ADP, relative to platelet-poor plasma (100% light transmittance). A lower MPA reflects stronger platelet inhibition, whereas a higher MPA reflects weaker inhibition.
Time Frame: Baseline, Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of aggregation
Arm/Group | 5 mg Prasugrel (Elderly) | 10 mg Prasugrel (Elderly) | 75 mg Clopidogrel (Elderly) | 5 mg Prasugrel (Non-Elderly) | 10 mg Prasugrel (Non-Elderly) | 75 mg Clopidogrel (Non-Elderly)
Number analyzed (Participants) | 72 | 70 | 71 | 78 | 79 | 79
percentage of aggregation
  Baseline | 79.10 (9.73) | 78.75 (9.53) | 79.11 (9.80) | 76.61 (8.07) | 76.61 (8.02) | 76.61 (8.02)
  Day 12 (n=71, 70, 70, 78, 79, 79) | 57.05 (13.98) | 45.54 (11.07) | 63.08 (13.73) | 56.83 (11.62) | 45.83 (11.82) | 59.09 (13.44)

ADVERSE EVENTS:
Arm/Group | 5 mg Prasugrel (Elderly) | 10 mg Prasugrel (Elderly) | 75 mg Clopidogrel (Elderly) | 5 mg Prasugrel (Non-Elderly) | 10 mg Prasugrel (Non-Elderly) | 75 mg Clopidogrel (Non-Elderly)
Serious Adverse Events (participants affected / at risk) | 0/73 | 2/71 | 2/72 | 0/79 | 2/82 | 0/79
Other Adverse Events (participants affected / at risk) | 20/73 | 31/71 | 25/72 | 23/79 | 39/82 | 23/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Prasugrel (Elderly) (N=73) | 10 mg Prasugrel (Elderly) (N=71) | 75 mg Clopidogrel (Elderly) (N=72) | 5 mg Prasugrel (Non-Elderly) (N=79) | 10 mg Prasugrel (Non-Elderly) (N=82) | 75 mg Clopidogrel (Non-Elderly) (N=79)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Prasugrel (Elderly) (N=73) | 10 mg Prasugrel (Elderly) (N=71) | 75 mg Clopidogrel (Elderly) (N=72) | 5 mg Prasugrel (Non-Elderly) (N=79) | 10 mg Prasugrel (Non-Elderly) (N=82) | 75 mg Clopidogrel (Non-Elderly) (N=79)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 4 (4)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 5 (6) | 9 (12) | 4 (9) | 1 (1) | 6 (6) | 4 (4)
Ear abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bleeding time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood creatinine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac enzymes increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (6) | 1 (1) | 2 (2) | 4 (6) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 9 (10) | 2 (4) | 5 (6) | 9 (10) | 3 (5)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days